CLINICAL TRIAL: NCT01717846
Title: In Vivo Effect on Orencia (Abatacept) on the Apoptosis of T Cells, B Cells and Antigen Presenting (APC) Cells in Rheumatoid Arthritis
Brief Title: Effect on Orencia (Abatacept) on the Apoptosis of T Cells, B Cells and APC Cells in Rheumatoid Arthritis
Acronym: RA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The PI has left UCLA and we do not plan to pursue this study.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-356; IM101-356 (Other: BMS)
Record Dates: First submitted 2012-10-24; First posted 2012-10-31 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Apoptotic DNA Damage; Rheumatoid Arthritis; T-cell Lymphocytosis
Keywords: Apoptosos; Rheumatoid Arthritis; T cells, B cells; DAS28; Clinical Disease activity Index; CDAI
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Orencia Group is for RA patients who have not received any other biologic treatment, including abatacept previously, and whose doctor has determined that it is appropriate to treat their RA with Abatacept. If you are in Group 1, you will receive the study drug, Abatacept, given in an intravenous (IV - injected into a vein) as well as subcutaneous form. Abatacept, given in an intravenous injection is approved by the FDA for the treatment of RA.
  Interventions: Drug: Group 1 or Orencia treated group
- Arm 2 or group 2 (Other): Arm 2 or Group 2 is for RA patients who are being treated wth non-biologic DMARDS who, with their doctor, have decided that they will not be receiving treatment with Abatacept in the next six months. These patients will not receive the study drug abatacept.
  Interventions: Other: Group 2 (DMARDS treated group)

INTERVENTIONS:
Drug: Group 1 or Orencia treated group — Group 1 subjects will be given subcutaneous abatacept, 125 mg once a week upto 6 months.
  Other Names: Abatacept
  Arms: Arm 1
Other: Group 2 (DMARDS treated group) — Arm 2 or Group 2 is for RA patients who are being treated wth non-biologic DMARDS who, with their doctor, have decided that they will not be receiving treatment with Abatacept in the next six months. These patients will not receive the study drug abatacept.
  Other Names: Arm 2 or group 2
  Arms: Arm 2 or group 2

SUMMARY:
This proposal will test the hypothesis that Orencia affects apoptosis and apoptosis related genes/biomarkers in vivo in rheumatoid arthritis (RA) patients.

DETAILED DESCRIPTION:
Orencia may regulate apoptosis and apoptosis related genes in vivo in rheumatoid arthritis (RA) patient's cells. To date, no studies have been performed to evaluate the effect of Orencia on apoptosis in RA patients.

Primary: To determine the effect of Abatacept in the apoptosis of T cells, B cells and antigen presenting cells (APC) in RA patients at baseline, 3 months and 6 months.

Secondary: To evaluate the association between the changes in apoptosis to changes in disease activity measures (DAS28/ESR) over 6 months of treatment with subcutaneous injection of abatacept.

ELIGIBILITY:
Inclusion Criteria:

1. Over age 18
2. Meeting ACR Criteria 1987 for RA diagnosis
3. Naïve to treatment with abatacept
4. Must be able to understand information in the Informed Consent

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Previous exposure to abatacept.
3. History of a concomitant autoimmune disease (eg. SLE, PsA etc.)
4. Patients with history of cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
To measure the change in apoptosis of T cells, B cells and antigen presenting (APC) cells in Rheumatoid Arthritis between the baseline, 3 months and at 6 months time points | Base line, 3 and 6 months
  To determine the effect of Abatacept in the apoptosis of T cells, B cells and antigen presenting cells (APC) in RA patients at baseline, 3 months and 6 months.

SECONDARY OUTCOMES:
To measure the change in disease activity score (DAS28) between the baseline, 3 months and 6 months time points | Baseline, 3 and 6 months
  To measure the changes in disease activity score joint count (DAS28/ESR)

OTHER OUTCOMES:
To measure the change in clinical disease activity index between base line, at 3 months and 6 months time points. | Baseline, 3 and 6 months
  To measure the Clinical Disease Activity Index (CDAI), and Health Assessment Questionnaire (HAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ram P Singh, MS, Ph.D., Principal Investigator — University of California at Los Angeles, UCLA; Mihaela Taylor, MD, Study Director — University of California at Los Angeles (UCLA)
Locations (1):
- Univerity of California at Los Angeles, Los Angeles, California, United States